CLINICAL TRIAL: NCT04629313
Title: Usak University Faculty of Dentistry
Brief Title: GCF Levels of IL-1Beta, MIP-1 Alfa and G-CSF in Gingivitis and Stage I-II-III-IV Periodontitis Patients
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Ahu Dikilitaş, Principal investigator, Uşak University
Other Study IDs: UsakU6
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Periodontitis
Keywords: periodontal disease; periodontitis; cytokines
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- periodontal disease group: Gingivitis: BOP score of 10% or greater and PD≤3mm with no attachment or radiographic bone loss.
  SI Periodontitis: interdental AL of 1-2 mm, PD≤4 mm and no tooth loss SII Periodontitis: interdental AL of 3-4 mm, PD≤5 mm and no tooth loss SIII Periodontitis: interdental AL ≥5 mm, PD≥6 mm SIV Periodontitis: interdental AL ≥5 mm teeth, radiographic bone lose extending to middle or apical third of the root,
- periodontal healthy group: consisted of individuals with clinically healthy gingiva

SUMMARY:
Periodontal diseases are chronic diseases that occur as a result of a violation of the balance between microbial dental plaque and the host response. Gingivitis is a disease characterized by inflammation of the gums that occurs in one or more areas without loss of attachments.1 in periodontitis, an inflammatory event that begins in the gum along with gingivitis spreads to the periodontal ligament, alveolar bone and soft tissues that support the tooth, causing the destruction of these structures.2 Cytokines are low molecular weight proteins that participate in the initial and active stages of inflammation and immunity. In periodontal disease pathogenesis, cytokine response has been reported to play a very critical role in determining disease progression.3 IL-1beta, MIP-1alfa and G-CSF are key cytokines in chronic inflammatory diseases and have the potential to initiate bone loss and tissue destruction seen in periodontal disease.4the purpose of this study; it is to determine the degree of inflammation and periodontal destruction by determining the levels of IL-1beta, MIP-1alfa, G-CSF cytokines in the gum groove fluid of periodontal healthy and diseased individuals.

DETAILED DESCRIPTION:
Plaque index (PI), gingival index (GI), presence of bleeding on probing (BOP), pocket depth (PD) and clinical attachment level (CAL) were used After clinical evaluation, individuals were divided into 6 groups Healthy control groups, gingivitis groups, Stage I groups, Stage II groups, Stage III groups and Stage IV groups GCF samples were collected after clinical periodontal measurement. GCF was obtained using strips of filter paper Kolmogorov-Smirnov and Shapiro Wilk's tests used

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of periodontal diseases
* Individuals must have 16 permanent teeth in their mouth

Exclusion Criteria:

* Diabetes
* İmmunological diseases

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals who have periodontal disease will be selected
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Measurement of IL-1Beta, G-CSF, MIP-1alfa levels in GCF | GCF samples were collected in the morning hours 24-48 hours after clinical periodontal measurement. GCF was obtained using strips of filter paper† from the buccal part of an interproximal region.
  Measurement of GCF samples

CONTACTS AND LOCATIONS:
Overall Officials: ahu dikilitaş, Principal Investigator — University of Usak; fatih karaaslan, Study Chair — University of Usak; umut yiğit, Study Chair — University of Usak; esra özge aydın, Study Chair — University of Usak; Abdullah seçkin ertuğrul, Study Director — University of Usak
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)